# Strong Families Start at Home/ Familias Fuertes Comienza en Casa Full Protocol for Data Collection, Processing and Management

# A Home-based Video and Motivational Interviewing Intervention to Improve Preschoolers Diet Quality and Parent

Protocol Revision History Version Number: 1 Version Date:02/26/2021





| Study Team Roster | 2 |
|---|---|
| Participating WIC Sites | 3 |
| Study Abstract | 3 |
| Study Objectives | 4 |
| Overview of Study Timeline and Evaluation | 5 |
| Recruitment | 6 |
| Screening, Eligibility and Enrollment: | 9 |
| Possible Questions that may come up during Recruitment/Enrollment | 10 |
| Home Visitation Guide | 11 |
| Interview Guide | 13 |
| Overview of data collection visit Introduction Script for Data Collection Team Interviewer Administered Questionnaire Forms to be Completed Anthropometrics Height: For the child: Weight: | 13<br>15<br>13<br>16<br>17<br>17<br>17 |
| Video Set Up | 20 |
| Schedule recall & First Home Visit | 21 |
| Potential Questions/Scenarios During BL Visit | 18 |
| Second Dietary Recall & Randomization | 24 |
| Data Management & QA | 26 |
| Coding and Feedback CEBQ Coding Feedback | 27<br>27<br>30 |



# Study Team Roster

| Alison Tovar | PI | alison_tovar@uri.edu<br>4018749855 |
|---|---|---|
| Patricia Risica | Co-I | patricia_risica@brown.edu |
| Kim Gans | Co-I | Kim.Gans@chip.uconn.edu |
| Karen McCurdy | Co-I | kmccurdy@uri.edu |
| Ernestine Jenning | CHW supervision, MI training, and adherence | ernestine_jennings@brown.edu |
| Katelyn Fox | RA/ Project manager<br>Recruitment calls<br>In home data collection | katelyn fox@uri.edu<br>401-787-0821- personal<br>401-545-9105 - study |
| Andrea Ramirez | RA Recruitment calls In home data collection Video coding | andrea_ramirez@uri.edu<br>401-441-4812 |
| Amy Moore | RA<br>PRN | amy_moore@uri.edu |
| Maggi Samson | RA<br>Video coding | margaret_samson@my.uri.edu |
| Adam Brice | UGRA Phone 24 hour recalls NDSR data management | adam_brice@my.uri.edu |
| Ivone Sical | UGRA In home data collection NDSR data management | ivone_sical@my.uri.edu<br>401-500-9449 |
| Haley Blanchette | JWU Intern | hblanchette01@jwu.edu |
| Rachel | UGRA | |
| Patricia Castillo | CHW | 401-771-5018 |
| Yesicca Cranshaw | CHW | 401-300-2258 |
| Heidi Samayoa | CHW | 401-248-5008 |
| Rede Reyes | Data Collection | 401-835-7254 |
| Elka Arredondo | | elvarredondom@gmail.com<br>(401) 569-6616 |



# Participating WIC Sites

| Meeting Street/St Josephs | Megan Sheehy | msheehy@meetingstreet.org, |
|---|---|---|
| Tri County | Isabella Fiore | isabellefiore8@gmail.com<br>ifiore@westelmwood.org |

# Study Abstract

There is an urgent need to create effective interventions to help parents establish a healthy diet among their children early in life, especially among low-income and ethnically diverse families. U.S. children eat too little fruits and vegetables and whole grains, and too many energy dense foods, dietary behaviors associated with increased morbidity from cardiovascular diseases. Contributing to this poor diet is consuming foods outside the home, having unhealthy foods available in the home and lack of home-prepared meals. Parents play a key role in shaping their child's diet and best practices suggest that parents should involve children in food preparation, offer, model and encourage a variety of healthy foods. In addition, while parents help to shape food preferences, not all children respond in the same way and certain appetitive traits, such as satiety responsiveness (sensitivity to internal satiety signals), food responsiveness (sensitivity to external food cues), and enjoyment of food may help explain some of these differences. Prior interventions among preschool aged children to improve their diet have not used a holistic approach that fully targets the home food environment, by focusing on food quality, food preparation, and positive feeding practices while acknowledging a child's appetitive traits. This proposal will build upon pre-pilot work to develop and pilot-test the feasibility, acceptability and preliminary efficacy of a novel home-based intervention with low-income ethnically diverse families of preschool children to inform a future fully powered randomized controlled trial. The proposed 6month intervention, will include 3 monthly home visits by a community health worker (CHW) trained in motivational interviewing, that include in-home cooking demos. In between visits, parents will receive tailored text-messages 2x/wk. and monthly mailed tailored materials. During the last 3 months CHW phone calls will replace the home visits. The intervention will be tailored for individual families based on the child's appetitive traits.



The aims are as follows: **Aim 1.** To conduct focus groups with 40 ethnically diverse parents of preschoolers to inform the development of and adaptation of the intervention components; **Aim 2.** To conduct a pilot RCT with 60 parent-child pairs (30 intervention/30 control) to determine the feasibility and acceptability of the enhanced intervention and determine the preliminary efficacy on child diet quality, feeding practices and availability of healthy foods in the home. The proposed research will lay the groundwork for a larger RCT to educate, support, motivate, and empower low-income parents to prepare healthy meals and use healthy feeding practices, which will improve children's diets and ultimately their health.

# Study Objectives

Aim 1: To conduct a pilot randomized controlled trial with 60 parent-child pairs (30 intervention/30 control) from ethnically diverse, low-income families with preschoolers to:

Aim 1.1: Determine the feasibility and acceptability of the enhanced intervention. Aim 1.2 Determine the preliminary efficacy of the enhanced intervention on changes in children's diet quality (primary outcome) and parental feeding practices and availability of healthy foods in the home (secondary outcomes) and calculate effect sizes for a future randomized controlled trial (RCT).

We hypothesize that the intervention will be feasible and acceptable to parents and that parent-child pairs randomized to the intervention condition will demonstrate greater improvements in the outcomes after six months compared to the comparison condition (attention control of a school readiness intervention).

Exploratory aim: Explore how parents' skills, perceived competence and intrinsic motivation are related to changes in children's diet quality and parental feeding practices.

# Overview of Study Timeline and Evaluation

Data collectors will be involved primarily with recruitment, enrollment and data collection at baseline and 6 month follow up. All data collection and tracking will occur via RedCap



45 minutes

# Software. Each data collector will have their own username and password to enter data into RedCap.



Please view this video on the Basics of Redcap Data Entry

45-minutes

https://redcap.vanderbilt.edu/consortium/videoplayer.php?video=data\_entry\_overview\_02.mp4&referer=redcap.uri.edu&title=Overview%20of%20Basic%20Data%20Entry

6- month

45 minutes

45-minutes

Recruitment



Overview of Recruitment Plan: The goal is to recruit a total of 60 parent-child dyads. In order to do this we will use a variety of methods to reach low-income diverse participants in the community. The first will be via WIC nutritionists who have been CITI certified and can provide us with names and numbers of interested participants. If a WIC nutritionist has not been CITI certified they are not allowed to provide us with this information. NOTE: If you speak to someone who would like to gather names and numbers of interested parents, please speak to Katelyn Fox (see contact) and we can provide them with information on how to become CITI certified. We will also be placing flyers around the community including childcare centers, WIC offices, community centers, libraries etc. Research Assistants & Hilda Castillo will also be doing individual outreach in the community to recruit participants.

**Recruitment via WIC nutritionist:** WIC nutritionists will provide study flyer and use the following script to describe the study to parents of children ages 2-5 years old.

# **Information Script for WIC Nutritionist**

I would like to tell you about a study being led by Dr. Alison Tovar from the University of Rhode Island (*WIC Nutritionist shows flyer to participant*). This study is being done to help improve children's wellness and development and is for parents who have a child between the ages of 2-5 years of age. Parents will participate in one of two groups: a group to help families make mealtimes easier or a group to help children get ready to read. As part of the six-month program, you will be working with a support coach, who will come to your home for three home visits, call you over the phone for three calls and text messages. At the end of the program you can receive up to \$150 for participating. If you think you might be interested, I can write down your name and number and someone from the study will call you and check to see if you are eligible to participate. Would you be interested in learning more about this program and should I write down your name?

<u>If client says yes, then respond:</u> Great! I will be giving them your name and number and they will be following up with you over the phone in the next couple of days.

<u>If client says no, then respond:</u> No problem, thank you for listening.

Please note that the project manager, will obtain names and contact information from WIC nutritionist weekly and store in secure excel file 'SFSH Recruitment' on the CNCOP team drive.



**In-person Recruitment by Research Assistants**: Study staff will recruit at the following locations (WIC offices, child care centers, summer kick off events). RA will provide flyer and use the following script to describe the study to potential participants. The script can be found in the eligibility form on Redcap.

**Information Script for Recruiter** 

Are you interested in hearing about a program to help improve children's wellness and development and is for children ages 2-5 years? If caregiver says yes

I would like to tell you about a study being led by Dr. Alison Tovar from the University of Rhode Island. This study is being done for parents who have a child between the ages of 2-5 years of age. Parents will participate in one of two groups: a group to help families make mealtimes easier or a group to help children get ready to read. As part of the six-month program, you will be working with a support coach, who will come to your home for three home visits, call you over the phone for three phone calls and text messages. At the end of the program you can receive up to \$150 for participating.

Would you be interested in finding out if you are eligible for this program? If client says yes, then respond: Great, do you have 5 minutes to see find out if you are eligible to participate? If yes, then proceed to screening and enrollment in Redcap. Fill out recruitment contact information form & give to project manager to enter data into 'SFSH Recruitment' spreadsheet

If no, say, **Ok, when would be a good time to call you back to find out if you are eligible?** Write down the date/time to call back.

If client says not right now, then respond: No problem, we are going to be recruiting over the next six months, do you think you would like us to call you back at another time?

If client says yes, then respond: Great! We can take down your name and number and call you at a later date.

If client says No, I am just not interested, then respond: No problem, thank you so much for your time, we appreciate you listening to us.



#### **Covid Recruitment**

RA will share a study flyer via text message, email, or social media and use the following script to describe the study to potential participants. The script can be found in the eligibility form on Redcap.

# **Information Script for Recruiter**

Are you interested in hearing about a program to help improve children's wellness and development and is for children ages 2-5 years? If caregiver says yes

I would like to tell you about a study being led by Dr. Alison Tovar from the University of Rhode Island. This study is being done for parents who have a child between the ages of 2-5 years of age. Parents will participate in one of two groups: a group to help families make mealtimes easier or a group to help children get ready to read. As part of the six-month program, you will be working with a support coach, who will video chat with you for three visits, call you over the phone for three phone calls and text messages. At the end of the program you can receive up to \$150 for participating.

Would you be interested in finding out if you are eligible for this program? If client says yes, then respond: Great, do you have 5 minutes to see find out if you are eligible to participate? If yes, then proceed to screening and enrollment in Redcap. Fill out recruitment contact information form & give to project manager to enter data into 'SFSH Recruitment' spreadsheet

If no, say, **Ok, when would be a good time to call you back to find out if you are eligible?** Write down the date/time to call back.

If client says not right now, then respond: No problem, we are going to be recruiting over the next six months, do you think you would like us to call you back at another time?

If client says yes, then respond: Great! We can take down your name and number and call you at a later date.

If client says No, I am just not interested, then respond: No problem, thank you so much for your time, we appreciate you listening to us.



# Screening, Eligibility and Enrollment:

- 1. Access 'SFSH Recruitment' in CNCOP team drive for contact information
- 2. Contact weekly x 4 weeks, document all calls in 'SFSH Recruitment'
- 3. Either in person or over the phone when screening: Begin Redcap Data Collection
  - a. In Person: Log into Redcap app>Choose project based on preferred language>
  - b. Over the phone : Log into online Redcap project. ADD/EDIT RECORDS>ADD A NEW RECORD > RECRUITMENT > ENROLLMENT
  - c. Information Script for Recruiter
    Hello, my name is [name of RA] with the University of Rhode Island.
    You spoke to someone [date of recruitment] at [location of recruitment]
    about our study and mentioned that you may be interested. As a
    reminder, we are comparing two programs to improve children's
    health and wellbeing, one that focuses on making healthy mealtimes
    easier and one that focuses on reading and preparing for school. If
    you choose to participate, each parent and their child will be
    "randomized" into one of the two groups. This means that you are
    put into a group by chance, like a lottery or by

As part of the six-month program, you will work with a support coach and get three home visits, three phone calls and text messages. For the healthy mealtime group you would also do a cooking activity in your home with a culinary student from Johnson & Wales University. At the beginning and end of the program we would ask you to fill out some surveys and we would measure height and weight of you and your child. You will be given up to \$150 for participating. Would you be interested in finding out if you are eligible for this

program?

If client says yes, then respond: Great! Proceed to eligibility questions in Redcap & Open SFSH Google calendar to schedule BL visit

\*Note use google calendar first to schedule based on data collection team availability. BL Assessment is entered afterward into redcap using year-month-day format.

If client says no, then respond: No problem, thank you for listening.

4. If participant does not answer the phone

flipping a coin.

a. Information Script for Recruiter

Hello, my name is [name of RA] with the University of Rhode Island. You spoke to someone [date of recruitment] at [location of recruitment] about our study and mentioned that you may be interested. We are comparing two programs to improve children's health and wellbeing, one that focuses on making healthy mealtimes easier and one that



focuses on reading and preparing for school. As part of the sixmonth program, you will get three home visits, three phone calls and text messages and at the end of the program you can receive up to \$150 for participating. You will also receive a text and email regarding the study. If you are interested in participating in the study you can call us back at 401-542-9105 or respond to the email from strongfamilies@etal.uri.edu

#### 5. Text

- a. Hi, this is [name of RA] at the University of Rhode Island. We want to know if you are interested in participating in our study to help improve children's health and well being.
- b. Text flyer image.

#### 6. Email

a. Hi, this is [name of RA] at the University of Rhode Island. We want to know if you are interested in participating in our study to help improve children's health and well being. We are comparing two programs to improve children's health and wellbeing, one that focuses on making healthy mealtimes easier and one that focuses on reading and preparing for school. If you choose to participate, each parent and their child will be "randomized" into one of the two groups. This means that you are put into a group by chance, like a lottery or by flipping a coin.

As part of the six-month program, you will get three home visits, three phone calls and text messages and at the end of the program you can receive up to \$150 for participating. You will also receive a text and email regarding the study. If you are interested in participating in the study you can call us back at 401-542-9105 or respond to the email from <a href="mailto:strongfamilies@etal.uri.edu">strongfamilies@etal.uri.edu</a>

- b. Email flyer image.
- 7. Project manager assigns and notifies data collection team of baseline visit once scheduled.

Possible Questions that may come up during Recruitment/Enrollment

**Q.** They want to participate but they want to choose what group they are in. **Response:** We are so excited that you are interested in participating. Because this is a research study we want to make sure that the group you fall into is random or by flipping a coin and unfortunately I cannot control that. The good news is that both groups will be working closely with a support coach and receiving important materials for your child's health and development. Once the study is over, if you are interested, we would be happy to share the materials from the program you did not receive.



**Q**. Their child has allergies to foods.

**Response**: Unless their child has a severe allergy, they may still participate.

**Q** What is a diagnosed feeding disorder?

**Response**: A diagnosis from a doctor or other medical provider (such as a dietitian, speech language pathologist or occupational therapist) that severely impacts how you feed your child. Children with a feeding disorder may have had weight loss, nutritional deficiencies, need for nutritional supplements or problems with functioning.

**Q** Can multiple children participate.

**Response**: The study will focus on one child between the ages 2-5 that the parent chooses for data collection purposes but the intervention material can and should be applied as a family so that all family members may benefit.

NOTE: If other questions come up and you are not sure, please contact Katelyn Fox, Andrea Ramirez or Alison Tovar so that we can help you answer these questions and also add to our protocol.

Baseline Data Collection: Now that participants have been enrolled in the study, we will need to consent them and collect the baseline data. A reminder text / call for baseline visit will be sent via Mosio.

Data collection team confirm & prepare for baseline visit.

- 1. I-Pad (check that I-pad is charged)
  - a. Note download participants record prior to visit while on wireless by logging into redcap app using your pin then select MyProjects>HomeVisitingR34Intervention (select correct language)>refresh setup and data (click proceed to clear project from i-pad)>get partial set of data> select records needed>download checked records>
- Charger
- 3. Consent forms
- 4. Paper survey copies
- 5. Color copy of Townsend measure to show participant during interview



- 6. Stadiometer
- 7. Height adjustment ruler
- 8. Scale
- 9. NDSR Laptop
  - a. Note set up record prior to home entry so that you are ready to begin dietary recall as soon as the participant completes the consent process.Include:
    - i. Participant ID
    - ii. Child date of birth
    - iii. Gender
    - iv. Date of visit
    - v. Visit number (1 for home baseline, 2 for phone baseline, 3 for home follow up, 4 for phone follow up)
    - vi. Interviewer ID- Your initials
- 10. Charger
- 11.2 food amount booklets
- 12. NDSR notebook
- 13. measuring spoons/cups
- 14. food models
- 15. Incentive (\$35)
- 16. Coloring & crayons for kids
- 17. Disinfectant wipes
- 18. Antibacterial hand gel
- 19. Tripod & instructions for google drive & video recording

Covid Baseline Data Collection: Now that participants have been enrolled in the study, we will need to consent them and collect the baseline data.

Following Enrollment in the study the research team will mail package including:

- 1. One copy of the consent form in the preferred language.
- 2. Food amounts booklet
- 3. Instructions for sending the home video
- 4. Sheet with survey responses
- 5. Tripod
- 6. Magnets

Data collection team confirm & prepare for baseline visit.

- 20. I-Pad (check that I-pad is charged)
  - a. Note download participants record prior to visit while on wireless by logging into redcap app using your pin then select MyProjects>HomeVisitingR34Intervention (select correct language)>refresh setup and data (click proceed to clear project



# from i-pad)>get partial set of data> select records needed>download checked records>

#### 21. Charger

#### Home Visitation Guide

# Remember to:

- Ensure that you are dressed appropriately, you are entering their home as a
  research professional. Avoid clothing such as halter / tube tops, bare midriff,
  short skirts or dresses, see through or ripped clothing, or clothing that displays
  inappropriate messages or pictures. Pants/skirt and a shirt or dress are
  appropriate options.
- Be respectful of the home, follow the participants lead on where they would like the interview to take place and ask permission before placing belongings anywhere. If the participant is unsure about where to meet, you can let them know that you will be asking them questions, so if possible a quiet place would be great.
- 3. Avoid using the families restroom.

#### Safety:

- 1. Stay alert entering neighborhoods, parking, and walking
- 2. Identify safe areas (i.e. restaurants, telephones, rest rooms, police stations)
- 3. Leave jewelry at home
- 4. Leave purse at office or trunk
- 5. Carry necessary cash, keys, study badge and driver's license on person
- 6. If at anypoint you feel unsafe, remove yourself from the situation
- 7. Travel in pairs when possible
- 8. Trust your instincts
- 9. Take universal precautions by washing hands before/after visit

#### Interview Guide

- 1. Make sure that your are thoroughly prepared prior to your visit. Ensure you have all materials and have practiced the interview so that you are comfortable and confident with the material.
- 2. Establish rapport with the participant. Present in a confident and friendly manner. Remember how you introduce the study and how you answer questions will help the participants feel more comfortable and willing to participate.
  - a. Establish trust. Follow the script to ensure that participants know who you are, that you are working for the University of Rhode Island, and why we are conducting this research.



- b. Personalize the interaction. Ask what they would like to be called and what they call their child. Try to use their names throughout the interview.
- c. Listen actively- make eye contact, let the person know that you are listening for example by nodding/ using "mmhm" and be patient, allowing them to complete statements without interruption. Ask for clarification if necessary.
- d. Show empathy by putting yourself in the other person's shoes and validating their concern, ask for clarification when necessary, explain steps you will take to address their concerns, and provide rationale for what you are asking them to do. See "Potential Questions" for examples of how to respond to common concerns.
- 3. Collect accurate and reliable data; this requires that every participant hears exactly the same questions read in exactly the same way.
- 4. Remember that you are there to ask for and record respondent's answers, not to influence or advise them in any way.
- 5. Always remain neutral in your words and manner. Never express criticism, surprise, approval or disapproval of the questions you ask or of the answers respondents give.
- 6. Ask all questions in a simple straightforward way. If you feel uncomfortable asking certain questions, such as about food security, practice them repeatedly until you are more comfortable stating them in a matter of fact way.
- 7. Ask every question as written, do not simplify. If a participant asks for an explanation for a word or part of a question refers to "Possible Questions that may come up" for responses. If a question comes up during an interview please let Katelyn Fox know so that standard response can be added to protocol if needed.
- 8. Discourage unrelated conversation. Maintain a businesslike attitude and acknowledge answers with comments such as "I see" or "OK". If you must interrupt do so politely, such as "that sounds very interesting, but what I need to ask is... " or "I see what you mean, but let me repeat that last question"
- 9. If a participant appears uncomfortable because of a personal question or does not want to answer take time to reassure the responded that he/she may speak freely, restate confidential nature of the interview and if the participant does not wish to answer the question take note in the comment section in Redcap.
- 10. Remember that it is best **not to know** if they are in the intervention or control group. If at follow-up data collection, the participants tells you what group they are in, do not assume that this is correct and most importantly do not as the best to your ability let this influence how you collect the data.
- 11. Remember you do not want to rush through data collection, obtaining as accurate data is possible is critical to the success of the project. Having said that



it is also important to not overextend your stay and be efficient in collecting the data.

Overview of data collection visit

Introduction Script for Data Collection Team

Hello, my name is [name of RA's] with the University of Rhode Island. You spoke to someone [date of enrollment] to set up our visit today. This is [name of 2nd RA] they will be helping me today. First I will review the study and you will sign what is called an informed consent to make sure that you agree to participate. If at any time you have questions or concerns you may ask me at any time. We will then ask you some survey questions. This visit should take about 1 hour to complete. At the end of our visit, I will be explaining what the next steps of the program will be as well as setting up your first visit with your support coach. I will also be providing you with your first gift card. Do you have any questions before we begin?

\*COVID- confirm that family has received baseline packet including copy of the consent form, food amounts booklet, magnet, instructions for taking home video and tripod

#### Consent

Participants will fill out parental consent form in their preferred language. Explain consent to participant describing the study and what to expect in the next 6 months. Signing the consent is a very important time to ensure that the participant knows and understands what they study is about. Make sure correct participant ID is written on the consent form in the top right corner.

#### Covid-Consent

Participants will have a copy of the consent form in their preferred language. Explain consent to participant describing the study and what to expect in the next 6 months. Verbally ask for consent for each portion (participation, video, and child participation)

### 24-hr Dietary Recall

Introduction to Dietary Recall

First we will collect some information on what your child ate yesterday. Here is a booklet that helps us estimate amounts of foods and beverages your child consumed along with some measuring cups and spoons, we will use this a little later.

Follow prompts in NDSR for conducting 5-pass dietary recall.



Upon completion of the dietary recall the second data collector will begin the interviewer administered questionnaires. While survey is being completed complete first QA pass and set up stadiometer and scale for anthropometric measurements. This way you are able to ask any necessary clarifying questions prior to leaving the home.

#### Interviewer Administered Questionnaire

Surveys will be completed in RedCap: The surveys will be interviewer administered. Remember to read the questions slowly and clearly and remind the participant that you are always happy to read the question again if they have concerns. Remind them that you are not looking for a "right" answer and that we are not judging them, we are simply learning from them and looking for them to be as open and honest as possible with their answers.

To complete surveys enter Redcap App with your PIN>collect data>select participant> select baseline assessment>demographics (after each form select status unverified then select save and go to the next instrument)

Forms to be Completed

Demographics

Feeding questions

Child Eating Behavior Questionnaire (CEBQ)

Household chaos

Basic Psychological Needs Satisfaction and Frustration (BPNSF)

14-item Diet Assessment Parent

Healthy Kids (For this questionnaire please show the participant the printed color copy while you ask them the questions)

Reading Readiness Checklist

Self-regulation scale

Perceived competence scale

Home food environment & photo of kitchen/ cooking space for visit

\*\* note if over 1.5 hours for visit do not complete home food environment.



# Anthropometrics (Not Collected During COVID)

Anthropometrics will be obtained on both the child and the parent. Recommend measuring the parent first then the child.

# Height:

The stadiometer is used to measure stature.

Height adjustment ruler: A 15-centimeter (cm) plastic ruler is used to correct stature measurements when participants hair styles that interfere with the stadiometer headpiece placement, or when they are unwilling to remove their shoes.

- 1. Have the parent stand erect on the floorboard of the stadiometer with his or her back to the vertical backboard of the stadiometer. Make sure that the weight of the participant is evenly distributed on both feet.
- 2. The heels of the feet are placed together with both heels touching the base of the vertical board. Place the feet pointed slightly outward at a 60 degree angle.
- 3. If the participant has knock knees, the feet are separated so that the inside of the knees are in contact but not overlapping.
- 4. The buttocks, scapulae, and head are positioned in contact with the vertical backboard. It may not be possible for some children and most adults to place their heels, buttocks, scapulae and the posterior aspect of the head against the backboard while maintaining normal stature. In that case participant should be positioned so that only the heels and buttocks are in contact with the vertical board, and the body is positioned vertically above the waist.
- 5. The arms hang freely by the sides of the trunk with palms facing the thighs.
- 6. The adult is asked to inhale deeply and to stand fully erect without altering the position of the heels.
- 7. The head is maintained in the Frankfort Horizontal Plane position while the examiner lowers the horizontal bar snugly to the crown of the head with sufficient pressure to compress the hair.
- 8. Hair ornaments, buns, braids, etc. must be removed to obtain an accurate measurement. The examiner needs to make sure that the hair of the participant does not obscure the scale.
- After the measurement is read from the by the examiner and recorded by the recorder to the nearest 0.1 cm. Repeat twice. Take a third measurement if the first two measurements are > 1 cm from each other

#### For the child:

1. Working with the caregiver, and kneeling in order to get down to the level of the child:



- 2. Help the child to stand on the baseboard with feet slightly apart.
- 3. The back of the head, shoulder blades, buttocks, calves, and heels should all touch the vertical board. This alignment may be impossible for an obese child, in which case, help the child to stand on the board with one or more contact points touching the board.
- 4. The trunk should be balanced over the waist, i.e., not leaning back or forward. Ask the mother to hold the child's knees and ankles to help keep the legs straight and feet flat, with heels and calves touching the vertical board.
- 5. Ask her to focus the child's attention, soothe the child as needed, and inform you if the child moves out of position.
- 6. Position the child's head so that a horizontal line from the ear canal to the lower border of the eye socket runs parallel to the baseboard. To keep the head in this position, hold the bridge between your thumb and forefinger over the child's chin. If necessary, push gently on the tummy to help the child stand to full height.
- 7. Still keeping the head in position, use your other hand to pull down the headboard to rest firmly on top of the head and compress the hair. Read the measurement and record the child's height in centimetres to the last completed 0.1 cm (0.1 cm = 1 mm) Repeat twice. Take a third measurement if the first two measurements are > 1 cm from each other





# Weight:

Digital scale (Seca 813)



- 1. Before beginning to weigh the participants, be sure that the scale is placed on a flat, hard, even surface. It should not be placed on a loose carpet or rug, but a firm carpet that is glued down is acceptable.
- 2. If a child is 2 years old or older and will stand still, weigh the child alone.
- 3. Ask the mother to help the child remove shoes and outer clothing. Talk with the child about the need to stand still. Communicate with the child in a sensitive, non-frightening way.
- 4. Turn on the scale. When the number 0.0 appears, the scale is ready.
- 5. Ask the child to stand in the middle of the scale, feet slightly apart, and to remain still until the weight appears on the display. Record the child's weight to the nearest 0.01 kg. If the child jumps on the scale or will not stand still, you will need to use the tared weighing procedure instead.

Weigh a child using tared weighing Check to see that the mother has removed her shoes. Ask the mother to stand in the middle of the scale, feet slightly apart, and remain still. The mother's clothing must not cover the display or solar panel. Remind her to stay on the scale even after her weight appears, until the child has been weighed in her arms. With the mother still on the scale and her weight displayed. Gently hand the child to the mother and ask her to remain still. Record this weight in the Recap. Be careful to read the numbers in the correct order (as though you were viewing while standing on the scale rather than upside-down). x2

Repeat twice. Take a third measurement if the first two measurements are > 0.1kg from each other

Video Set Up

Provide Tripod, set up google drive, and review instructions.

As part of the intervention we would like you to video record a time with you and your child at a meal if you are feeding your child group and a time when you read or tell stories if you are in the school readiness group. We will review



the video and provide some feedback on what is working well and tips to help you. In order to do this you can film it on your cell phone. Here is a tripod that you can put your phone in and set it up nearby your child [demonstrate]. In order for you to send us the video securely we are using whatsapp or an app called google drive. Do you use Whatsapp? If not, would prefer to download it or use the google platform? Do you have a google email? Would you be willing to set one up? Now we can get the google photo app. [Have participant set up google photo app in visit, if they have an android phone they may already have it]] I will share a folder with you [If access to the internet can create folder with participant number in visit]. Now you can upload the video to this folder (demonstrate).

# Covid Video Set Up

Parents should have received a tripod and instructions in the mail. Describe above and if possible offer to set up video chat to demonstrate if the family has any questions.

#### Schedule recall & First Home Visit

Just a reminder we are comparing two programs to improve children's health and wellbeing, one that focuses on making healthy mealtimes easier and one that focuses on reading and preparing for school. You and your child will be "randomized" into one of the two groups. This means that you are put into a group by chance, by flipping a coin. This will be decided after you complete the next call over the phone next week where we ask you similar questions to what we did today to find out what your child ate. Let's schedule the day for that call now.

# We would also like to take the time to schedule your first visit with the support coach.

Refer to support coach calendar/times that are available and offer those times. Google Calendar "Strong Families Start at Home Study" with window of 3 weeks from baseline visit +/- 4 days.

Enter date into redcap.

Let parents know they will receive a \$35 gift card & inform participants that they will receive an additional \$15 at their first home visit if they complete the 2nd phone call to ask them about what their child ate.

Ask preference for how they would like to receive gift card and include in notes section - can receive walmart (via email or mail) or target (via text, email, or mail).

Upon returning to the office, complete the following:



- Sync data to online project by RedCap app> my project (choose correct language project)> Send Data to Server
- 2) Scan and upload a copy of the consent into Redcap
- Confirm that all data was entered and synced. Review all dates and measurements for data entry errors. Change status of form from Unverified to complete.
- 4) Complete first QA pass
- 5) Return all materials to room 119.
- 6) If any questions came up during the data collection process please check as soon as possible with Katelyn/Alison about these issues.

Potential Questions/Scenarios During BL Visit

#### Consent

Potential concerns & responses

When addressing participants concerns or responses remember to show empathy by putting yourself in the other person's shoes and validating their concerns explain steps staff will take to minimize concern and provide rationale for what we are asking them to do.

Examples

"I don't think I would be comfortable with so my family meal/ reading"

Validate their concern and ask for clarification (Note in the statement above the parent does not explain why they would not be comfortable so you can't address their concern.)

You could say: "I understand you may feel uncomfortable recording your family. What are your concerns about this"?

They may say "I worry about privacy

Or

"I worry it will be embarrassing"

# Explain steps to address concern

"We understand that your family's privacy is extremely important. You will send us the video using an application. The study staff who review the video will not see your name or any identifying information. The videos will be stored in secure server. The only people that will see your video are yourself, the study staff, and the support coach who will come to your home, after 5 years the videos will be deleted" Or



"We understand that it may feel uncomfortable to film you and your child. The person reviewing the videos will not see your name or any identifying information The goal of the video is not to judge you or grade you on how well you interact with your child. We understand that children in this age range are very unpredictable and that is normal"

# Provide rationale for what you are asking them to do

"The reason we have you provide the video is so that we can see if watching and receiving feedback on family videos can help parents find ways to improve their children's health. We have tried something similar with other families and they found it very helpful.

Parents: "I'm not sure about someone coming into my home"

## Validate their concern and ask for clarification if necessary

Researcher: "We understand that having someone come to your home may be uncomfortable. Is there something specific that you are worried about?

They may say "How will I know who they are"

Or

"I worry they would judge our family"

Or

"I wouldn't be comfortable if it was a male"

## Explain steps to address concern

It is important to us that you feel comfortable and safe.

Study personnel will have a badge with the URI logo & their name printed on it. All study personnel are registered with our institutional review board, have completed several hours of training and have experience working in family's homes. Their role is to provide you information and help you set goals to improve your family's health not to judge you in anyway.

Or

We can ensure that you only have female personnel \*\* Please make a note of this in redcap and alert Katelyn so that all female data collection teams are assigned\*\*

# Provide rationale for what you are asking them to do



We are conducting a home-based study because we understand families are busier than ever and want to ensure everyone has access regardless of transportation or schedule.

# Demographics

Q. What is my race/ethnicity?

**Answer:** Remember that you can not identify race/ethnicity just by looking at a person. Provide the following explanation and allow the participant to identify themselves.:

# **Ethnicity**

**Hispanic or Latino** - A member of an ethnic group that traces its roots to 20 Spanish-speaking nations from Latin America and Spain itself.

#### Race

**White** – A person having origins in any of the original peoples of Europe, the Middle East, or North Africa.

**Black or African American** – A person having origins in any of the Black racial groups of Africa.

**American Indian or Alaska Native** – A person having origins in any of the original peoples of North and South America (including Central America) and who maintain tribal affiliation or community attachment.

**Asian** – A person having origins in any of the original peoples of the Far East, Southeast Asia, or the Indian subcontinent including, for example, Cambodia, China, India, Japan, Korea, Malaysia, Pakistan, the Philippine Islands, Thailand, and Vietnam.

**Native Hawaiian or Other Pacific Islander** – A person having origins in any of the original peoples of Hawaii, Guam, Samoa, or other Pacific Islands.

# Second Dietary Recall & Randomization

- 1. Project manager will notify phone call recall team when recalls are scheduled.
- 2. UGRA will log into redcap to obtain participant contact information & enter redcap form. Find participant record> event pre\_visit1> Second Recall



- 3. Fill out header section in NDSR prior to beginning recall
  - a. Participant ID
  - b. Child date of birth
  - c. Gender
  - d. Date of visit
  - e. Visit number (1 for home baseline, 2 for phone baseline, 3 for home follow up, 4 for phone follow up)
  - f. Interviewer ID- Your initials
- 4. If participant answers the phone.
  - a. RA will complete 5 pass dietary recall per NDSR protocol
- 5. After Foods have been entered into NDSR:
  - a. Notify participants that incentive will be given to them at their first home visit when the support coach comes(\$15).
  - b. Open randomization envelope and let participants know which group they are in and enter form in redcap
    - i. Remind participants of the video recording.

As part of this program we ask that you video record a time with your child. As you are in the (identify group assignment) we ask that you record a (meal with your child or a time that you read with your child). Do you have any questions about this? Do you remember how to use Google Photo to share your videos with us?

6. If participant does not answer the phone leave message & document call attempt in RedCap. Attempt x2 to get weekday weekend, if not 2 weekday.

Hello, my name is [name of RA] with the University of Rhode Island . I am calling to complete the last part of the interview so that we can begin the program.. Please give us a call back at 401-542-9105. After the interview you will be given your study group and you will also receive a second gift card for your time.

In the event that the second recall is not completed within two weeks of the baseline visit, the participants will then be randomized without completing that second recall. Since they have their home visit scheduled they will find out at that time.



# **Data Management**

NDSR Data Entry Rules & Assumptions

- 1. Follow NDSR training data entry rules (Appendix 15 of the NDSR manual) unless otherwise noted. Ensure that there are complete and <u>detailed</u> notes for any items entered. This includes documenting what the participants said their child ate, what was used to estimate portion sizes and any other relevant information
- If no recipe exists for a food item, if standard recipes in NDSR do not suffice, and participant knows the ingredients and amounts used create a user-recipe for the meal in NDSR.
  - a. If recipe quantities are available:
    - i. Create user recipes with the quantities and ingredients noted.
    - ii. Be sure to keep recipe name in original language
  - b. If recipe quantities are not available:
    - i. Follow NDSR "Mixed Foods" protocol follow the prompts on screen, and choose appropriate ingredient variables.
    - ii. If mixed foods are not appropriate, make substitution based on best, most similar available food item in NDSR.
    - iii. Priority note all recipes for review by CNCOP data management.
- QA of NDSR data entries Recall
  - a. Missing foods and substitutions protocol
    - i. Missing foods are considered a last resort if no appropriate substitution is available for your food product in NDSR. appropriate substitutions are determined by the following nutrient tolerances:

## **Nutrient tolerances per 100g of product**

| Calories | +/- 85.0 kcal |
|--------------------|---------------|
| Protein | +/- 5.00g |
| Total fat | +/- 2.50 g |
| Total carbohydrate | +/- 10.00g |
| Sodium | +/- 100.00 mg |

b. If the nutrient values of the closest food substitute **does not** fall within the nutrient tolerance per 100g, then the product will be considered a missing food.



- This will be determined after the 3rd QA pass usually by the lead RDN whether or not a MF is appropriate.
- Missing foods will be resolved via NCC (Nutrition Coordinating Center).
  - a. Submit a New Food request form (have nutrition facts for product available).
  - b. The missing foods client number for URI is: 679 ir University of Rhode Island.
- 4. Determine the appropriate substitution(s) for item(s) that are not found in NDSR.
  - a. Print the Nutrients per Food report.
    - i. NDSR R34 project >> Click on record ID that has the substitution>> Reports tab >> Nutrients per food.
  - b. Compare the nutrients of the substitution to the actual food product.
    - i. You will need to find the nutrition information from online or producer.

Coding and Feedback

CEBQ Coding

Export CEBQ data into SAS by clicking Data Exports, Reports, and Stats> Selected instruments and or events> CEBQ and Baseline> export raw data without labels

Score CEBQ using code title "CEBQ\_Score". Enter category into redcap.



- a) If CEBQ SR=1 then participant is "low satiety responsiveness"
- b) If CEBQ FF=1 then participant is "high food fussiness"
- c) If CEBQ FR=1 then participant is "high food responsiveness"

If participant is high in multiple traits, they will first get tailored information on the food fussiness, followed by satiety responsiveness and then food responsiveness.

```
CEBQ Score Code
data redcap.CEBQ;
SET redcap.CEBQ;
reverse cebg3= 6-cebg3 bigappetite;
reverse_cebq4= 6-cebq4_finishesquickly;
reverse CEBQ10= 6-cebq10 enjoystasting;
reverse CEBQ16= 6-cebq16 enjoysvariety;
reverse CEBQ32= 6-cebq32 interestedtasting;
Run:
data redcap.CEBQ;
set redcap.CEBQ;
CEBQ FF= (cebq7 refusesnew+reverse CEBQ10+reverse CEBQ16+
reverse CEBQ32+cebq35 moreslowly)/6;
CEBQ FR= (cebq12 alwaysasking+ cebq14 eattoomuch+ cebq19 mostofthetime+
cebg28 favoritefoods+cebg34 alwaysfood)/5;
CEBQ SR= (REVERSE CEBQ3+ cebg17 leavesfood+ cebg21 fullbefore+
cebq26 fulleasily+ cebq30 mealsnack)/ 5;
Run;
Data redcap.CEBQ;
set redcap.CEBQ;
if CEBQ SR<2.8 then low SR=1;
if CEBQ SR>=2.8 then low SR=0;
if cebq_sr=. then low sr=.;
if cebg FF>3 then high FF=1;
if cebq ff<=3 then high FF=0;
if cebq ff=. then high ff=.;
if cebq FR>2.8 then high FR=1;
if cebq FR<=2.8 then high FR=0;
if cebg fr=. then high FR=.;
run;
```

Enter results in Final Baseline Checklist form of Baseline Visit in Redcap.

Video Coding



Project manager will monitor study WhatsApp and Google account daily. When video is received video coding staff will be notified and sent video. Video should be coded within one week of receiving.

If video is not received within 1 week of randomization a text message will be generated to remind the participant.

If the video is not received within 2 weeks of randomization a phone call and text message will be sent to remind the participant and answer any questions they may have about the purpose of the video or how to record/send the video.

# Protocol for video coding:

- 1. Project manager will alert coders when a new video is uploaded to the server.
- Prior to watching the video, have Operational Definitions and Coding Tool readily accessible. While the coder will have the Operational Definitions available to them during the coding process, it is important that they are comfortable with identifying the different practices.
- 3. Watch video and fill out coding sheet. It is likely that the video may need to be paused multiple times while coding, and certain clips may need to be re-watched if the parental practices seem ambiguous. For further directions on when to code, refer to the directions on the top of the Operational Definitions sheet.
- 4. While watching the video, note if there is a specific interaction that stands out in a positive or negative way, or if a behavior occurs multiple times within a meal. If there is not a positive and negative clip that stands out, use best judgment to select a clip.
- 5. Follow below protocol to edit the video so it contains only the "positive" and "negative" clips.
- Fill out the CHW Feedback Sheet by writing a quick overall description of the meal at the top of the sheet. Mention anything that may be beneficial for the CHW to know about the meal (Remember that the CHW will not be viewing the full video).
- 7. Briefly describe what practice the video clip is showing.
- 8. Copy and paste the appropriate sample feedback. Modify as necessary so that feedback is specific to what is observed in the video, and upload to the CHW's folder on the Google Drive.
- 9. Go onto RedCap application, and copy the information from coding tool onto the "Video Coding" tab.



# Protocol for video editing using iMovie:

- 1. In order to edit the video with the positive and negative clip, import the entire video into iMovie.
- 2. Create a new project and name it StudyID\_VideoClips\_1 or StudyID\_VideoClips\_2.
- 3. When in the "My Media" tab of the "Projects" section, drag the clip to the bottom half of the screen (it should be a lighter gray than the top).
- 4. Trim the video so it only includes the desired positive clip by moving the bidirectional arrow cursor that will appear at the front and end of the clip.
- 5. Add a title slide that says "Clip 1" before the video clip. Find this by clicking the "Titles" tab, and dragging the desired title to the bottom half of the screen.
- 6. Repeat Step 5 to create a title slide that says "Clip 2" following the first positive video clip.
- 7. Repeat steps 3 and 4 to trim the clip to only include the desired negative video clip.
- 8. Export the video by going to the "File" tab, then "Share", then "File". The video clips will then be downloaded as a .mov

#### Feedback

Project manager will upload video clips, feedback form, and CEBQ trait into CHW google drive folders. If the participant does not complete the video sample video and feedback sheet will be provided.

CHW will be notified via email and text message when new materials are uploaded.

#### NDSR QA protocol

- 1. Open NDSR and select the project and the record.
- 2. Review the **Header** tab
  - Check to ensure that the record is entered into the correct project
  - Check the participant ID & DOB with redcap ID and DOB
  - Check the date of intake (typically the day before the date of entry).
  - Check the interviewer ID
  - Check the visit number (1 for home baseline, 2 for phone baseline, 3 for home follow up, 4 for phone follow up)
- 3. Review the **Food** tab.



- Review each food name for correctness. Visualize what is eaten.
- Review each amount. Visualize how much is eaten. Use the reference amount (in parenthesis) as another reality check.
- Use study approved amount estimation tools or ruler to "re-create" amounts.
- Are Food Amounts Booklet amounts entered correctly?
- Make sure Assembled Foods include a complete description of the food.
- Are all components of the food included? (e.g, bread for the sandwich)
- Are companion foods included? (e.g, spread for bread or toast, bread or rolls with a restaurant meal.
- Are amounts appropriately described and reasonable?
- o Is a rationale documented for unusually small or large portions?
- Do Missing Foods include complete descriptions of food and amount eaten?
- 4. Review the **Trailer** tab.
  - Read Notes for completeness and accuracy.
- 5. View the **Quick List**. Make sure foods entered correspond to the Quick List and account for all foods initially reported. Make notes for discrepancies.
- 6. Generate and review the **Nutrients per Food Report.** 
  - Check the gram weight for unusual amounts
    - 8 FO (fluid ounces of coffee) = 240g (beverages vary in density).
    - 6 FO of wine = 176g (6 oz = 170.10g).
    - $\blacksquare$  1 ½ cup of frosted cheerios = 35g (8 ounces = 227g = 6.075 cp).
    - 2 medium tomato slices = 40g (2 medium tomatoes = 123g)
    - 1 medium brownie = 2" x 2" = 40g
  - Other reference points include: 28g of cheese = 1oz; 454g of steak = 1 pound; 250g of chili = 1 cup.
  - Check individual food items that are >400kcal, >25g fat, >500g total weight.
- 7. Generate the Missing Foods and Missing DSAM Products List Reports
  - Select the sample project missing for the training project.
  - o From the Reports menu, select the Missing Foods List Report.
  - When asked if you would like to open the Missing Foods List Report or save it, select Open.

**Note:** This report opens as an excel file which can be formatted as desired. You may wish to document your QA decisions in an additional column on this report. It also may



be helpful to copy and paste the missing foods and decisions into a master list for use throughout your study.

- 8. Generate and Review the Food and QA Report
  - Highlight the project and Your Name W001 in NDSR.
  - From the Reports menu, select the Quality Assurance Reports > Foods QA
     Report
  - When asked if you would like to open the Foods QA Report or save it, select Open. As you review the report, highlight items on the spreadsheet that may need editing.
    - Check data for items that need to be fixed or require interviewer education.
    - Sort by **Note** field. Review priority notes. Look for items that require editing, research, or data entry decisions.
  - Highlight **Unit Selected** column and search for OZ. Verify that beverages are entered with FO instead OZ.
  - For larger data-sets sort by **Food ID** to place like items together to check for the amount errors.
- 9. Return to NC003 in your W001 project and make corrections to problems identified.
- 10. Generate a new **Foods QA Report**. Review Food Detail Notes.

**Note:** Use the **Record Search** to find a record during the QA report revi

## Data Backup

All data (Redcap & NDSR) will be exported and backed up each Friday on the teams external hard drive in folder StrongFamilies\_Backup. Please refer to NDSR Healthy Start protocol for more information on NDSR data entry and cleaning.

### Blinding

Data collectors will be blinded to what arm the participant is in. You will not know if they are in the intervention or control group.

# Completion/Final Evaluation

Final evaluations will be scheduled by the support coaches during their last visit. All data collection teams should have their availability entered in the google calendar Repeat all data collection procedures outlined above.



# Reporting Procedures

# Injury

In the event of any injury to the participant or to yourself, data collection staff should immediately report to supervisor, Katlyn Fox or Alison Tovar. In consultation with the project manager, PI and co-I, if appropriate, unexpected problems/outcomes should be reported on Appendix S – Event Reporting. Management staff to report to IRB

#### Child abuse

Please immediately report to supervisor (Katelyn Fox and Alison Tovar) if you have any concern that you have witnessed child abuse.

A report is required when:

- A person has reasonable cause to know or suspect that a child has been abused or neglected.
- "Any recent act or failure to act on the part of a parent or caretaker which results in death, serious physical or emotional harm, sexual abuse or exploitation"; or
- "An act or failure to act which presents an imminent risk of serious harm."

If you are not sure, please discuss with Katelyn or Alison and a decision can be made.

## Study Discontinuation

**Lost to Follow Up**. If a participant does not attend scheduled visit and team is unable to contact the participant protocol is to Contact by phone, text and email 2 x/week x 2 weeks.

**Expresses desire to discontinue study.** If a participant expresses desire to discontinue the study alert project manager. Thank them for participating and ask, if willing to share, the reason for discontinuation. Project manager will cancel all upcoming visits/ data collection time points.

Data will be kept for all participants who have been randomized prior to discontinuation and analyzed with intention to treat .



# Training

All data collectors

NDSR training binder

Quality control Metrics

Protocol deviations

Monitoring

**IRB** Review

# **Measures & Coding**

Feeding Question Sub-Scale & Coding

| FPI | Question | Variable<br>Name |
|---|---|---|
| Encourage Trying New Foods | | |
| Offer New Foods | I teach my child about new foods | fpi_teach |
| | I offer new foods at mealtime | fpi_offerm |
| | I offer new foods at snack | fpi offers |



| Encourage Exploration of<br>New Foods | I let my child explore new foods by smelling | fpi_explores |
|---|---|---|
| | I let my child explore new foods by licking or touching the food to his/her lips | fpi_explorel |
| | I let my child explore new foods by picking up and looking at the foods | fpi_lookfood |
| Urge Child to Eat New Foods (mean inter-item correlation = .33) | When I offer new foods, I have my child eat at least one bite | fpi_onebite |
| | I show my child how to try foods by taking a bite myself | fpi_bitemyself |
| | I have my child try a new food before he/she eats sweet foods | fpi_beforeswe<br>et |
| | If my child refused to eat a new food, or a food he/she does not like, I continue to offer that food | fpi_continue |
| Repeated Presentation of<br>New Foods | If my child does not eat a new food on one day, I offer it again on another day | fpi_offeragain |
| | If my child does not eat a new food on one day, I offer it again and prepare it in a different way on another day | fpi_offerprepa<br>re |
| | I offer foods for my child to try even if I don't like them myself | fpi_dontlike |
| Mealtime Structure | | |
| Family Meals | Our family regularly eats dinner together | fpi_dinnert |
| | Everyone if our family is expected to be home for dinner | fpi_homedinn<br>er |
| | People in our family feel strongly about eating dinner together | fpi_together |



| | People in our family sit in the same seats at every meal at home | fpi_samesit |
|---|---|---|
| Regular Timing of Meals and Snacks | We have routine times for meals at our house | fpi_routineme<br>al |
| | We have routine times for snacks at our house | fpi_routinesna<br>ck |
| | Having a routine time for children to eat is important | fpi_routine |
| Inconsistent Mealtimes | Adults in our house have separate mealtimes from children | fpi_adultm |
| | Dinnertime in our family is flexible. People eat whenever they can. | fpi_flexible |
| | In our family, there is little planning around dinnertime | fpi_pland |
| Indifferent Feeding | An effective way to get an upset child to quit crying is to feed him/her | fpi_crying |
| | My child can have juice when he/she asks for it | fpi_juice |
| | Children should be able to eat foods they want to for snacks | fpi_wantsnack<br>s |
| | I have bigger problems to worry about than which foods my child is eating | fpi_biggerpro<br>blem |
| Child Involvement in Food Preparation | My child helps me prepare new foods | fpi_helpprepa<br>re |
| | My child helps prepare part of the meal | fpi_preparem |
| | My child helps prepare his/her snacks | fpi_prepares |
| Parent Decides Portion<br>Sizes | I put food on my child's plate | fpi_childsplate |



| | I serve the right amount so that my child can eat enough | fpi_eatenough |
|---|---|---|
| | Are you responsible for the size of the portions your child receives? | fpi_portionsiz<br>e |
| | Are you responsible for how many helpings your child gets? | fpi_helpchild |
| Serves Measured Portions | I help my child use a tablespoon so that he or she knows how much food should go on the plate | fpi_spoon |
| | I measure portions for myself based on food packaging guidelines | fpi_portionm |
| | I measure portions for my child based on food packaging guidelines | fpi_portiongui<br>des |
| External Control | | |
| Pressure to Eat | If my child says "I'm not hungry," I try to get him/her to eat anyway | fpi_nothungry |
| | I have to be especially careful to make sure my child eats enough | fpi_careful |
| | My child should always eat all of the food on his/her plate | fpi_plate |
| | If I did not guide or regulate my child's eating, he/she would eat much less than he/she should | fpi_eatless |
| Restriction | I have to make sure that my child does not eat too many sweets | fpi_eatsweets |
| | I have to make sure that my child does not eat too many high fat foods | fpi_highfats |
| | If I did not guide or regulate my child's eating, he/she would eat too many junk foods | fpi_junkfood |
| Food as a Reward | I offer sweets to my child as a reward for good behavior | fpi_offersweet |



| | I offer my child his/her favorite foods as a reward for good behavior | fpi_favoritef |
|---|---|---|
| | A favorite food is an effective way to reward children | fpi_foodrewar<br>d |
| Responsiveness to Child's Fullness Cues | When my child resists eating, I ask him/her if he/she is hungry | fpi_resisteatin<br>g |
| | During mealtime I ask my child is his/her stomach is full | fpi_fullstomac<br>h |
| | During meals, I ask if my child is still hungry | fpi_hungryd |
| Monitoring | Do you keep track of the sweets that your child eats? | fpi_trackswee<br>ts |
| | Do you keep track of the snack foods that your child eats? | fpi_tracksnac<br>ks |
| | Do you keep track of the high fat foods that your child eats? | fpi_trackfat |



# Assumptions & Data Entry Rules

| Date Entered | Data Entry Form | Rule |
|---|---|---|
| 8/9/17 | NDSR | If meat is fried and option not available in NDSR (ie for sausage) assume that fat absorbed by the meat is 1.5% of the total weight of the meat. For example: If 85g sausage is fried in butter assume that 1.3 g of butter is absorbed (85g x 0.015=1.3g) |
| 8/9/17 | Demographic Form & Healthy<br>Kids Form | If given a range of times choose the mean. For example if reports bedtime is between 20:00 and 21:00 enter as 20:30. |
| 8/9/17 | Demographic Form<br>Ages of children in the home | Enter age as years. For example if parent reports child is 3 months enter as 0.25 years. |
| 8/9/17 | 14 Item Diet Screener | If parent reports 1 tsp of cream/butter/ margarine per day enter. If >1.5 tsp count enter as 1 x/week |
| 8/9/17 | Healthy Kids | Record fortified non-dairy milks as soy milk. |
| 8/9/17 | 14 Item Diet Screener | If eating red meat >3x/week enter 1 x/day. |
| 8/27/17 | NDSR | 1 bite of hamburger = 15 g (1/16th) |
| 9/3/19 | NDSR | Breastfeed unknown volume assume 2 oz per feeding https://jandonline.org/article/S 0002-8223(10)01481-1/pdf |



| 9/3/19 | NDSR | Every attempt to be made to quantify amount using FAB or measuring spoon/cup. However if only estimate provided is large serving spoon assume ½ cup. |
|---|---|---|
| 9/25 | NDSR | If supplement n/a in NDSR Katelyn or Andrea will find similar supplement in NDSR. Please enter all supplement details in notes section so that in the future we request the supplement if necessary. |
| 10/23 | NDSR | Dip with carrots is 1 Tbsp low fat ranch on CACFP menu |
| 11/13 | NDSR | For pizza eaten without crust subtract 1" from radius of wedge. If wedge size N/A decrease portion by 20%. |
| 2/26 | NDSR | ½ CP milk per 1 CP cereal |
| 08/21 | NDSR | 1TB of oatmeal per 8 FO for oatmeal drink |
| 08/25 | NDSR | If amount of water not provided, use amount from another day. |
| 8/31/20 | NDSR | Sugar on cereal (included oatmeal)= 1 TS sugar per 1 CP cereal |
| 9/2/2020 | NDSR | Medium slice pizza: 7 D (FAB) |
| 09/04/2020 | NDSR | For banana, a bite is an inch |
| 10/1/2020 | NDSR | 1 bite : 1 TB (M3)<br>1 sip: 1 FO |
| 10/1/2020 | NDSR | Dip from childcare menu:<br>dips, unknown type, unknown<br>if regular or fat-free |

